CLINICAL TRIAL: NCT05239767
Title: A Randomized Trial of NSAID Dosing Strategies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-13802
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Musculoskeletal Pain; Acute Pain
MeSH Terms: conditions — Musculoskeletal Pain; Acute Pain | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: NSAID will be masked. Acetaminophen or no acetaminophen will not
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Active Comparator): Ketorolac 20mg orally x 1
  Interventions: Drug: NSAID
- Ibuprofen (Active Comparator): Ibuprofen 800mg orally x 1
  Interventions: Drug: NSAID

INTERVENTIONS:
Drug: NSAID — We will administer oral NSAIDs

SUMMARY:
This study will compare the efficacy of two different non-steroidal anti-inflammatory drugs (NSAIDs) ketorolac and ibuprofen for people with acute moderate or severe musculoskeletal pain. The investigators will also determine whether taking acetaminophen prior to the NSAID impacts efficacy

ELIGIBILITY:
Inclusion Criteria:

* Acute musculoskeletal pain: Any pain attributable to muscles, bones, joints, tendons, ligaments or supporting structures, as determined by the clinical team, of 10 days duration or less. Prior to the onset of acute pain, patients cannot have experienced pain in the same body region during the prior six months
* Pain has to be described as moderate or severe, when the patient is asked if the pain is mild, moderate or severe in intensity

Exclusion Criteria:

* Contraindication to NSAIDs (allergy to NSAID or allergy to aspirin without history of tolerating NSAIDs, history of gastrointestinal bleeding, daily medication for gastritis or PUD, chronic kidney disease 2-5, heart failure)
* Contraindication to acetaminophen (hepatitis or cirrhosis)
* Use of an NSAID within the previous eight hours
* Use of acetaminophen within the previous eight hours
* Chronic pain, defined as any pain on >50% of days for at least 3 months prior to onset of acute pain
* Recurrent pain in the same body part as the presenting complaint

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 407 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Failure to achieve a minimum clinically important difference | Two hours
  Failure to improve by at least 1.3 points on a 0-10 pain scale

SECONDARY OUTCOMES:
0-10 pain score | One and two hours after medication administration
  Improvement on 0-10 pain
Ordinal pain scale | One and two hours after medication administration
  The investigators will determine the frequency of obtaining pain levels of "mild" and "none" on a scale of "severe", "moderate', "mild", or "none"
Epigastric pain | Two hours after medication administration
  Participants will be asked if the medication caused "stomach pain". Response options are "no", "a little", "a lot"

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No